CLINICAL TRIAL: NCT04700085
Title: Reverse Innovation in Western Health Care: the ReMotion Prosthetic Knee.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 837_ReMotion_Knee
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Knee
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial design
Masking Description: Participants and researcher could not be blinded as participants performed a training session with the ReMotion Knee (one of the conditions) and the prosthetic knee type was visible to both.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReMotion Knee (Experimental): The ReMotion Knee (mechanical prosthetic knee type) was used during measurements
  Interventions: Device: ReMotion Knee
- Current prosthetic knee (No Intervention): The participant's current prosthetic knee was used during measurements

INTERVENTIONS:
Device: ReMotion Knee — The ReMotion Knee is a prosthetic knee mostly used in low-income countries. It has been approved according to the ISO 10328 standards and has received the CE Mark.
  Arms: ReMotion Knee

SUMMARY:
Ambulatory mobility and function are important aspects in the quality of life of people with lower limb amputations and prostheses. Regaining mobility is often challenging, especially for patients with transfemoral, or above-knee, amputations. In the past decades, new types of knee prosthetics have entered the market. The standard care in Europe and the US at this moment is the mechanical, or non-microprocessor controlled, knee (NMPK). While the production costs of these NMPK's are lower than those of the MPK's (microprocessor controlled knee), consumer prices still reach up to $5000. Recently, the ReMotion Knee ($80) was developed as a new and affordable alternative to the currently available mechanical knees. The ReMotion Knee is mostly used in low-income countries, but has now been approved according to the ISO 10328 standards and has received the CE Mark. This knee could be a more affordable alternative for the prosthetic knees used in high-income countries, thereby decreasing health related costs within the amputation population. However, research on patient's functional abilities and personal experiences with the knee is very limited and has not been investigated within more developed countries. Therefore, the objective of this study is to compare the ReMotion Knee and the current prosthetic knee of patients with a transfemoral amputation or knee-exarticulation in terms of functional mobility, balance, and experienced walking comfort, balance trust, fatigue and performance of the knee. it is expected that the ReMotion Knee will perform slightly worse than the participants' current prosthetic knees.

DETAILED DESCRIPTION:
The primary aim of healthcare organizations is to optimize the quality of life of their patients while keeping a good balance between quality and costs. More advanced medical technologies are constantly being developed to improve quality of life. However, these technologies also lead to rising healthcare costs in high-income countries. Cost pressures from medical innovations, along with the ageing population form a substantial threat to the long-term sustainability of healthcare systems in high-income countries. Reverse innovations (products or ideas originally designed for use in low-income countries that are 'upgraded' and implemented in high-income countries) provide an opportunity to restrain the rising healthcare costs in high-income countries. These products are often low-priced, easy to use, and designed to function and survive in extreme and unpredictable conditions. However, low-income country of origin products are still generally perceived as less reliable and safe and they are rarely researched as an alternative to the current standard of care within the medical sector.

The field of lower limb prosthetics is a typical example of a medical field with unceasing technological developments, accompanied by rising expenses. With the rising incidence of lower-limb amputations and the rising prosthetic prices, the costs of prosthetics care will keep increasing. Reverse innovation could play an essential role in controlling the costs of prosthetic care in the upcoming decades. However, research on new, lower-priced alternative prostheses for use in high-income countries is very scarce and deserves more attention. An example of a potential reverse innovation for the prosthetics market is the ReMotion knee: an $80 mechanical knee recently designed by D-Rev (San Francisco, CA, USA) for use in low-income countries. The ReMotion Knee has a polycentric design and a lifespan of about 3-5 years, comparable to other mechanical knees, but does not include a pneumatic or hydraulic system. It is easy to use, provides patients with a basic functional mobility, and is low priced, especially compared to the standard care mechanical knees ranging between $1000 and $4000 in the Netherlands. The ReMotion Knee could in this new way propose an opportunity to greatly reduce healthcare costs among amputees in high-income countries. So far there is no research available on health outcomes with the ReMotion Knee other than overall user satisfaction, and it has never been evaluated as an alternative prosthetic knee for use in high-income countries.

This study aims to evaluate the ReMotion Knee as a potential reverse innovation and provide insight in the value of reverse innovation. To this end, the ReMotion Knee was compared with currently used and comparable mechanical prosthetics knees in high-income countries. The knees were evaluated based on the most important health outcomes for people with a lower-limb amputation: functional mobility, walking comfort, balance and trust in balance. Furthermore, experienced fatigue and performance with the knees were examined. As the ReMotion Knee has less features advanced features than most polycentric prosthetic knees currently used, it was expected that all would be slightly lower with the ReMotion Knee.

ELIGIBILITY:
Inclusion Criteria:

* Medicare Functional Classification Level (MFCL) 2 or 3 (most probable users of the ReMotion Knee)
* at least one year since amputation
* currently using a polycentric mechanical prosthetic knee.

Exclusion Criteria:

* stump pain that increases with activity
* a hip flexion contracture > 20 degrees
* inability to stand and walk for thirty minutes
* weight >80kg (weight limit of the ReMotion Knee)
* a prosthetic socket connection that did not fit the ReMotion Knee
* an osseointegrated prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
L-test | 5 minutes
  Measure for functional mobility

SECONDARY OUTCOMES:
Four Square Step Test (FSST) | 5 minutes
  Measure for presicion stepping
Berg Balance Scale (BBS) | 15 minutes
  Measure for static balance
Weight distribution during static stance | 2 minutes
  Measure for static balance
Modified Emory Functional Amputation Profile (mEFAP) | 5 minutes
  Measure for functional mobility
Experienced walking comfort | On average, after 30 minutes and after 90 minutes
  Experienced walking comfort is measured with a visual analog scale (VAS) of 10 centimeters (lowest score is 0, highest score is 10).
Experienced trust in balance | On average, after 30 minutes and after 90 minutes
  Experienced trust in balance is measured with a visual analog scale (VAS) of 10 centimeters (lowest score is 0, highest score is 10).
Experienced performance of the knee | On average, after 30 minutes and after 90 minutes
  Experienced performance of the knee is measured with a visual analog scale (VAS) of 10 centimeters (lowest score is 0, highest score is 10).
Experienced fatigue | On average, after 30 minutes and after 90 minutes
  Experienced fatigue is measured with a visual analog scale (VAS) of 10 centimeters (lowest score is 0, highest score is 10).

CONTACTS AND LOCATIONS:
Overall Officials: Noël LW Keijsers, PhD, Study Chair — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No